CLINICAL TRIAL: NCT05162352
Title: Donafenib Combined With Sintilimab for Advanced HCC: a Single-arm, Single-center, Prospective Study
Brief Title: Donafenib Plus Sintilimab for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-08
Record Dates: First submitted 2021-12-01; First posted 2021-12-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Donafenib; Sintilimab; TKI; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Donafenib+sintilimab (Experimental): Donafenib combined with sitilimab.
  Interventions: Drug: Donafenib+sintilimab

INTERVENTIONS:
Drug: Donafenib+sintilimab — Part 1 (Safety Run-in): donafenib 200mg P.O. BID and sintilimab 200mg I.V. for a 21-days cycle.
  Part 2: donafenib at the recommended phase 2 dose determined from Part 1 and sintilimab 200mg I.V. Q3W.
  Donafenib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Sintilimab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Patients will be allowed to have donafenib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

SUMMARY:
This study will evaluate the efficacy and safety of donafenib combined with sintilimab in patients with advanced hepatocellullar carcinoma (HCC).

DETAILED DESCRIPTION:
This is a Phase II study to evaluate the efficacy and safety of donafenib combined with sintilimab in patients with advanced HCC.

30 subjects with advanced HCC (Barcelona-Clinic- Liver-Cancer [BCLC] stage C, or China liver cancer staging [CNLC] IIIa/IIIb) will be enrolled in the study.

Part 1 (Safety Run-in): 6 patients will receive donafenib 200mg P.O. BID and sintilimab 200mg I.V. for a 21-day cycle.

Part 2: patients will receive donafenib at the recommended phase 2 dose determined from Part 1 and sintilimab 200mg I.V. Q3W.

Donafenib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Sintilimab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Patients will be allowed to have donafenib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC (BCLC stage C or CNLC IIIa/IIIb ) with diagnosis confirmed by histology/cytology or clinically
* Patients who have Tumor recurrence after surgical resection or ablation are allowed to be included
* Patients who previously received local treatment, such as transcatheter arterial chemoembolization, transcatheter arterial embolization and radiotherapy, are allowed to be included
* At least one measurable lesion
* Child-Pugh score ≤7
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and hematologic function
* Life expectancy of at least 3 months

Exclusion Criteria:

* Diffuse HCC
* Macrovascular invasion involving the main trunk or inferior vena cava
* Central nervous system metastasis
* History of malignancy other than HCC
* Esophageal and/or gastric varices bleeding within 3 months prior to initiation of study treatment
* Uncontrolled ascites
* History of hepatic encephalopathy
* Patients who received prior systemic therapy (chemotherapy, targeted therapy or immunotherapy) or hepatic arterial infusion chemotherapy (HAIC) for HCC
* History of organ and cell transplantation
* Active severe infection; use of antibiotics within 2 weeks prior to injection of sintilimab
* Autoimmune disease or immune deficiency
* Severe organ (heart, kidney) dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-04 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by investigators according to modified Response Evalutaion Criteria in Solid Tumors (mRECIST). | 18 months
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events (AEs) | 18 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), AE of special interest (AESI), serious adverse event (SAE), assessed by NCI CTCAE v5.0.
PFS assessed by investigators according to Response Evalutaion Criteria in Solid Tumors (RECIST) v1.1 | 18 months
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Objective response rate (ORR) assessed by investigators according to mRECIST. | 18 months
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Disease control rate (DCR) assessed by investigators according to mRECIST. | 18 months
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD).
ORR assessed by investigators according to RECIST 1.1. | 18 months
  The percentage of patients who had a best overall tumor response rating of CR or PR.
DCR assessed by investigators according to RECIST 1.1. | 18 months
  The percentage of patients who had a tumor response rating of CR, PR, or SD.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Dr., Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hong X, Guo Y, Shi W, Zhu K, Liang L, Lin L, Chen Y, Zhou J, Huang J, Huang J, Wu Y, Huang W, Cai M. Donafenib combined with sintilimab for advanced hepatocellular carcinoma: a single arm phase II trial. BMC Cancer. 2025 Feb 5;25(1):205. doi: 10.1186/s12885-025-13605-2. PMID 39910472